CLINICAL TRIAL: NCT03613714
Title: Innovation in Postpartum Care for Women With Hypertensive Disorders of Pregnancy: A Randomized Trial of Home- Versus Office-Based Blood Pressure Monitoring
Brief Title: Innovation in Postpartum Care for Women With Hypertensive Disorders of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18-0995
Record Dates: First submitted 2018-07-25; First posted 2018-08-03 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Hypertension in Pregnancy; Hypertension, Pregnancy-Induced; Postpartum Preeclampsia; Blood Pressure Disorders
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): At-home blood pressure monitoring at 2-5 days post-discharge from the hospital using a digital blood pressure cuff. Participants will receive text message reminders to check blood pressure. Contacted by clinic staff to review blood pressure log.
  Interventions: Other: At-home Blood Pressure Monitoring
- Usual Care (No Intervention): Blood pressure monitoring assessment will be done at 2-5 days post-discharge in the office. Participants will be given high blood pressure information hand-outs and instructed to follow-up in obstetric clinic for blood pressure check within 5 days after discharge from the hospital.

INTERVENTIONS:
Other: At-home Blood Pressure Monitoring — Participants will use over-the-counter digital monitor to measure blood pressure and pulse rate at home. Automatically averages the last 3 readings taken over 10 minutes.
  Other Names: Digital Blood Pressure monitoring cuff
  Arms: Intervention Group

SUMMARY:
Hypertensive disorders of pregnancy (HDP) affect up to 10% of mother-infant dyads and account for 7.4% of cases of maternal mortality in the United States. Prompt recognition and treatment of hypertension remain one of the key features of management of mothers affected by these conditions. Up to 41% of severe morbidity and mortality from HDP occurs after 48 hours postpartum, as postpartum blood pressures tend to peak 3-6 days after birth. For these reasons, early postpartum follow-up is recommended for women diagnosed with HDP, in the form of blood pressure (BP) evaluation by a health care provider at 7-10 days postpartum (2-5 days post-discharge from maternity care). However, barriers to follow-up limit mothers' ability to adhere to this recommendation. A potential alternative to in-office evaluation is at-home BP monitoring. At-home BP monitoring is a novel, affordable method to empower, educate, and engage postpartum women affected by HDP. Within the obstetric (OB) population, pilot studies have demonstrated the feasibility and acceptability of remote BP monitoring. Hence, the purpose of this randomized trial is to empower postpartum women affected by HDP and cared for at North Carolina Women's Hospital to perform at-home BP monitoring with the aid of digital technology.

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy (HDP) affect up to 10% of mother-infant dyads and account for 7.4% of cases of maternal mortality in the United States. Prompt recognition and treatment of hypertension remain one of the key features of management of mothers affected by these conditions. Improving recognition and treatment is of particular importance given that maternal mortality rates continue to rise in the United States. Moreover, mothers affected by HDP are at increased risk of long-term morbidity, such as cardiovascular disease, atherosclerosis, and persistent hypertension outside of pregnancy. Therefore, it is critical to recognize hypertension throughout maternity care, including in the postpartum period.

The postpartum period is a time of major challenges for the new mother and considerable physiologic changes that place the new mother at increased risk of adverse events. For a postpartum woman with a diagnosis of a HDP, the risk of complications extends beyond discharge from maternity care: up to 41% of severe morbidity and mortality from HDP occurs after 48 hours postpartum, as postpartum blood pressures tend to peak 3-6 days after birth. For these reasons, the American College of Obstetricians and Gynecologists (ACOG) and the National Partnership for Maternal Safety recommend early postpartum follow-up for women diagnosed with HDP, in the form of blood pressure (BP) evaluation by a health care provider at 7-10 days postpartum. However, barriers to follow-up, including childcare arrangements, transportation access, and recovery from delivery, limit mothers' ability to adhere to this recommended in-office follow-up. Indeed, attendance at postpartum follow-up visits is poor and reflects significant disparities.

A potential alternative to in-office evaluation is at-home blood pressure (BP) monitoring. At-home BP monitoring is a novel, affordable method to empower, educate, and engage postpartum women affected by HDP. This approach is not in widespread use in the US, despite the American Heart Association indicating that home BP monitoring is recommended for all people with high blood pressure. Within the obstetric population, pilot studies have demonstrated the feasibility and acceptability of remote BP monitoring. However, a randomized trial of postpartum at-home BP monitoring compared with office-based follow-up is lacking.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Diagnosis of a hypertensive disorder of pregnancy (HDP)
* Chronic hypertension requiring medications

Exclusion Criteria:

* Less than 18 years or older than 60 years
* No access to cellular telephone
* Chronic hypertension not on medications during pregnancy or postpartum
* No diagnosis of HDP
* Upper arm circumference < 9 inches or > 17 inches
* Incarcerated mother
* The woman requires a 1-week postpartum in-office visit for other medical reason unrelated to the diagnosis of hypertensive disorder of pregnancy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who undergo a BP evaluation by clinic staff at 2-5 days post-discharge | 2-5 Days Post Hospital Discharge
  BP evaluation will be counted if performed by clinic staff via telephone or in person if documented in the medical record.

SECONDARY OUTCOMES:
Percentage of participants readmitted for inpatient management of severe hypertension within 2 weeks of delivery | 2 weeks from delivery
Percentage of participants readmitted within 2 weeks of delivery | 2 weeks of delivery
  Readmission, regardless of indication, within 2 weeks of delivery
Percentage of participants requiring OB triage evaluation for severe hypertension within 2 weeks of delivery | 2 weeks after delivery
Percentage of participants with severe hypertension who present to OB triage or Emergency Department for recommended same-day evaluation | Within 24 hours after BP evaluation
  Includes those diagnosed with severe hypertension in the office or through phone follow-up
Percentage of attendance to recommended 4-to-6-week postpartum visit | Up to 6 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Angelica Glover, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the results will be shared
Time Frame: Beginning 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data must have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB) and execute a data use/sharing agreement with UNC.